CLINICAL TRIAL: NCT04583228
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of HLX71 in Healthy Adult Subjects
Brief Title: Evaluate the Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of HLX71 (Recombinant Human Angiotensin-converting Enzyme 2-Fc Fusion Protein for COVID-19) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hengenix Biotech Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: HLX71-001US-253460
Record Dates: First submitted 2020-09-25; First posted 2020-10-12 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The investigators plan to enroll 8 subjects in each sequence, of which 2 receive intravenous injection of placebo and 6 receive intravenous injection of IP. Subjects are allocated in two groups randomly.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A total of 32 subjects were randomized in a double blind fashion with 24 subjects receiving active drug and 8 subjects receiving placebo. Eight subjects were randomized in each dose cohort at a 3:1 ratio, with 6 subjects receiving active drug and 2 subjects receiving placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sequence 1 (Experimental): Random allocation to HLX71 1 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 8 receive intravenous injections of the HLX71.
  Interventions: Drug: HLX71; Other: Placebo
- Sequence 2 (Experimental): Random allocation to HLX71 3 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 8 receive intravenous injections of the HLX71.
  Interventions: Drug: HLX71; Other: Placebo
- Sequence 3 (Experimental): Random allocation to HLX71 10 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 8 receive intravenous injections of the HLX71.
  Interventions: Drug: HLX71; Other: Placebo
- Sequence 4 (Experimental): Random allocation to HLX71 15 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 8 receive intravenous injections of the HLX71.
  Interventions: Drug: HLX71; Other: Placebo

INTERVENTIONS:
Drug: HLX71 — Single-dose, intravenous infusion
  Other Names: Recombinant Human Angiotensin-Converting Enzyme 2-Fc Fusion Protein
Other: Placebo — Single-dose, intravenous infusion

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of HLX71 in Healthy Adult Subjects

DETAILED DESCRIPTION:
A randomized, double-blind, single-dose by intravenous administration, placebo-controlled, dose escalation, first-in-human study is proposed to evaluate the safety, tolerability, pharmacodynamics, pharmacokinetics and immunogenicity of HLX71 in healthy subjects. Investigators plan to enroll 10 subjects in each of the 4 dose cohorts at 2.5 mg/kg, 5 mg/ kg, 10 mg/kg and 15 mg/kg, of which 2 receive intravenous injections of placebo and 8 receive intravenous injections of the investigational product (IP). A total of 40 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with voluntary signing of the informed consent form (ICF), and capable of understanding and following the requirements.
* Healthy males or females aged ≥ 18 and < 65 years at the time of signing the ICF.
* Body weight ≥ 50.0 kg and < 100.0 kg, and body mass index (BMI) ≥ 18.5 kg/m2 and < 30.0 kg/m2.
* The subject is in good health as determined by the Investigator according to medical history, physical examination, vital signs, 12-lead ECG, chest X-ray, and laboratory tests (hematology, serum chemistry, C-reactive protein, thyroid function, coagulation, etiology, urinalysis).
* No plan of pregnancy and being willing to use continuous effective contraception for subjects (including partner) from informed consent to 6 months after administration of investigational product, see Appendix 1 for the specific contraceptive measures.

Exclusion Criteria:

* Subjects with the lab-confirmed medical history of COVID-19, including SARS-CoV-2 determined by reverse transcription-polymerase chain reaction (RT-PCR) or positive specific antibody IgM or IgG against serum SARS-CoV-2.
* Subjects with the novel onset of pyrexia/cough/shortness of breath/diarrhea or history of contact with confirmed COVID-19 individuals within the 14 days before randomization.
* Pneumonia or active tuberculosis (TB) indicated by chest X-Ray, or abnormal and clinically significant as judged by the Investigator.
* Abnormal blood pressure or pulse rate: systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg, SBP ≤ 90 mmHg or DBP < 60 mmHg, pulse rate < 50 beats /min or > 100 beats/min at screening and clinically significant as judged by the Investigator.
* Clinically significant 12-lead ECG abnormalities, or QTcF interval > 450 msec at screening, or history of clinically significant ECG abnormalities, which may increase the risk to the subject as judged by the Investigator.
* Use of monoclonal antibodies or fusion proteins within 6 months before screening.
* Subjects with previous exposure to vaccines in 3 months before screening, or who plans to receive vaccination during the study period or in 3 months after the study.
* History of allergy to any monoclonal antibody, fusion protein, biological product, protein product, or ingredient of the IP.
* Family history of cardiovascular disease, history of atherosclerosis, presence of chronic obstructive pulmonary disease (COPD), cirrhosis, cardiovascular disease, or any condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being.
* History of blood loss or blood donation (including blood component donation) ≥ 400 mL, or reception of blood transfusion within 3 months prior to screening; blood loss or donation (including blood component donation) ≥ 200 mL within 1 month prior to screening.
* Previous surgery within 2 months before screening, or scheduled surgery during the study.
* Previous administration of any investigational drugs/comparators in clinical trials within 3 0 days or remaining in the elimination period of the drug (within 5 half-lives) before screening, or still in the follow-up period of a certain clinical study.
* Use of prescribed drugs, over-the-counter (OTC) drugs, or herbal medicines (excluding vitamins and mineral supplements) within 14 days before screening.
* History of alcohol abuse or intake of excessive alcohol in the past 6 months (15 unit of alcohol per week: 1 unit = 285 mL beer, or 25 mL liquor, or 100 mL wine), or alcohol breath test positive, or unwilling/unable to quit alcohol drinking during the study.
* Subjects who smoke ≥ 5 cigarettes per day or are positive in tobacco screening , or those who are unwilling/unable to quit nicotine intake during the study.
* Positive for hepatitis B surface antigen (HbsAg), hepatitis C virus antibody (anti-HCV), human immunodeficiency virus antibody (anti-HIV) antibody, treponema pallidumparticle agglutination test (TPPA) or Tuberculosis (TB) quantiferon at screening.
* Positive β-Human Chorionic Gonadotropin (β-HCG) or breastfeeding female subjects.
* History of narcotics abuse or addiction, or positive drug screening.
* Other conditions unsuitable for participation in the study determined by the Investigator, such as potential compliance issues, inability to complete all tests and evaluations required in the protocol, and uncontrolled psychiatric or mental illnesses.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, serious adverse event and infusion-related reactions as assessed by CTCAE v5.0 | up to 28 days
The proportion of subjects undergoing DLT events in each dose cohorts during the DLT observation period | Days 1 to 7

SECONDARY OUTCOMES:
PK parameters-Peak concentration | Pre-infusion, immediately post-infusion(0 hours), 1, 2.5, 4, 10, 24 hours after end of infusion and on days 3, 4, 6, 8, 10, 12, 15, 18, 22 and 29
PK parameters-Time to peak | Pre-infusion, immediately post-infusion(0 hours), 1, 2.5, 4, 10, 24 hours after end of infusion and on days 3, 4, 6, 8, 10, 12, 15, 18, 22 and 29
PK parameters-Areas under the concentration-time curves | Pre-infusion, immediately post-infusion(0 hours), 1, 2.5, 4, 10, 24 hours after end of infusion and on days 3, 4, 6, 8, 10, 12, 15, 18, 22 and 29
PK parameters-Terminal elimination rate constant | Pre-infusion, immediately post-infusion(0 hours), 1, 2.5, 4, 10, 24 hours after end of infusion and on days 3, 4, 6, 8, 10, 12, 15, 18, 22 and 29
PK parameters-Elimination half-life | Pre-infusion, immediately post-infusion(0 hours), 1, 2.5, 4, 10, 24 hours after end of infusion and on days 3, 4, 6, 8, 10, 12, 15, 18, 22 and 29
PK parameters-Clearance (CL) | Pre-infusion, immediately post-infusion(0 hours), 1, 2.5, 4, 10, 24 hours after end of infusion and on days 3, 4, 6, 8, 10, 12, 15, 18, 22 and 29
PK parameters-Volume of distribution | Pre-infusion, immediately post-infusion(0 hours), 1, 2.5, 4, 10, 24 hours after end of infusion and on days 3, 4, 6, 8, 10, 12, 15, 18, 22 and 29
The concentration-time curves of plasma Ang1-10 | Pre infusion, immediately post-infusion(0 hours), 1, 4, 10, 24 hours after end of infusion and on days 3, 8, 15 and 29
The concentration-time curves of plasma Ang1-9 | Pre infusion, immediately post-infusion(0 hours), 1, 4, 10, 24 hours after end of infusion and on days 3, 8, 15 and 29
The concentration-time curves of plasma Ang1-8 | Pre infusion, immediately post-infusion(0 hours), 1, 4, 10, 24 hours after end of infusion and on days 3, 8, 15 and 29
The concentration-time curves of plasma Ang1-7 | Pre infusion, immediately post-infusion(0 hours), 1, 4, 10, 24 hours after end of infusion and on days 3, 8, 15 and 29
The concentration-time curves of plasma aldosterone | Pre infusion, immediately post-infusion(0 hours), 1, 4, 10, 24 hours after end of infusion and on days 3, 8, 15 and 29
ADA positive rate | Day 15 and 29
NAb positive rate | Day 15 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, MD, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No